CLINICAL TRIAL: NCT02770807
Title: Multi-center, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Effects of Intra-Erythrocyte Dexamethasone Sodium Phosphate on Neurological Symptoms in Patients With Ataxia Telangiectasia
Brief Title: Intra-Erythrocyte Dexamethasone Sodium Phosphate in Ataxia Telangiectasia Patients
Acronym: ATTeST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Quince Therapeutics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IEDAT-02-2015; 2015-005241-31 (EudraCT Number)
Record Dates: First submitted 2016-05-02; First posted 2016-05-12 (Estimated); Results first posted 2024-05-09 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Nervous System Disease; Genetic Syndrome
Keywords: Ataxia Teleangiectasia; AT; EryDex system; Dexamethasone; Dexamethasone sodium phosphate
MeSH Terms: conditions — Nervous System Diseases; Genetic Diseases, Inborn

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The Sponsor, Investigator, site staff, and patients were not aware of the treatment assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EryDex Low Dose DSP (Experimental): EDS-EP dose range of ~5-10 mg DSP/infusion. This study treatment was to be administered by IV infusion once per month for 12 consecutive months (6 months Initial Treatment Period + 6 months Extension Treatment Period). Each patient underwent a 30-day Screening Period, during which any previous treatments with other corticosteroid compounds were withdrawn (washout from previous treatment).
  Other Names:
  EryDex System end product Low dose DSP
  Interventions: Drug: EryDex Low dose DSP
- EryDex High Dose DSP (Experimental): EDS-EP dose range of ~14-22 mg DSP/infusion. This study treatment was to be administered by IV infusion once per month for 12 consecutive months (6 months Initial Treatment Period + 6 months Extension Treatment Period). Each patient underwent a 30-day Screening Period, during which any previous treatments with other corticosteroid compounds were withdrawn (washout from previous treatment).
  Other Names:
  EryDex System end product High dose DSP
  Interventions: Drug: EryDex High dose DSP
- Placebo (Placebo Comparator): Patients were treated with autologous erythrocytes prepared with the EDS process using a placebo solution. Placebo was to be administered by IV infusion once per month for 12 consecutive months (6 months Initial Treatment Period + 6 months Extension Treatment Period).
  Each patient underwent a 30-day Screening Period, during which any previous treatments with other corticosteroid compounds were withdrawn (washout from previous treatment).
  Interventions: Drug: Pooled Placebo

INTERVENTIONS:
Drug: EryDex Low dose DSP — EDS-EP dose range of ~5-10 mg DSP/infusion
  Other Names: EryDex System end product
  Arms: EryDex Low Dose DSP
Drug: EryDex High dose DSP — EDS-EP dose range of ~14-22 mg DSP/infusion
  Other Names: EryDex System end product
  Arms: EryDex High Dose DSP
Drug: Pooled Placebo — EDS processed autologous erythrocytes using a sodium chloride [NaCl] solution.
  Other Names: Placebo EDS infusion
  Arms: Placebo

SUMMARY:
Objectives:

The objective of study was to evaluate the safety and the efficacy of EryDex (Dexamethasone sodium phosphate encapsulated in autologous erythrocytes, using the EryDex System - EDS) at two dose levels (low dose and high dose DSP/infusion), compared to placebo, on Neurological Symptoms in Patients With Ataxia Telangiectasia.

Initial Double-Blind Treatment Period (0 to 6 Months)

Primary Efficacy Objective:

• Evaluate the effect of EryDex at two dose levels (low dose and high dose DSP/infusion), compared to placebo, on central nervous system (CNS) symptoms measured by the change in the Modified International Cooperative Ataxia Rating Scale (mICARS) from baseline to Month 6 (Visit 9) in patients with ataxia telangiectasia (A-T).

Secondary Efficacy Objectives:

* Evaluate the effect of EryDex, compared to placebo, on the Clinical Global Impression of Change (CGI-C) in patients with A-T from baseline to Month 6 (Visit 9).
* Evaluate the effect of EryDex, compared to placebo, on measures of Clinical Global Impression of Severity (CGI-S; structured) in patients with A-T from baseline to Month 6 (Visit 9)
* Evaluate the effect of EryDex, compared to placebo, on measures of Adaptive behavior measures in patients with A-T by the Vineland Adaptive Behavior Scales (VABS) from baseline to Month 6 (Visit 9).

Safety Objectives:

• Evaluate the safety and tolerability of two non-overlapping doses of EryDex, compared to placebo, in patients with A-T over the 12-month double-blind study duration.

Extension Treatment Period (6-12 Months):

Primary Objective:

• Evaluate the efficacy of EryDex at two dose levels (low dose and high dose DSP/infusion) compared to placebo, in treating CNS symptoms in A-T patients during longer-term treatment (up to 12 months), as measured by the mICARS.

Secondary Objectives:

* Evaluate the longer-term (up to 12 months) safety and tolerability of EryDex in A-T patients.
* Compare the effects of EryDex on the CGI-C and CGI-S (structured), VABS, and QoL using the EQ-5D-5L scale.

DETAILED DESCRIPTION:
This was an international, multi-center, one-year, randomized, prospective, double-blind, placebo-controlled, phase III study.

This study was divided into three periods: Screening (Days -30 to -1), 6-month Initial Treatment Period (Months 1-6; Visits 1-9), and 6-month Extension Treatment Period (Months 7-12; Visits 10-15).

A total of 175 patients, of the 180 planned, met all selection criteria at baseline, and were randomized in a 1:1:1 fashion to one of the two EDS-EP dose levels or placebo.

These patients were randomly assigned to receive one of the two doses of EDS-EP or placebo, as follows:

* Group 1: EDS-EP dose range of ~5-10 mg DSP/infusion (low dose), 59 pts
* Group 2: EDS-EP dose range of ~14-22 mg DSP/infusion (high dose), 57 pts
* Group 3: Placebo EDS infusion, 59 pts

The initial 6-month treatment period was considered complete when the endpoint assessment (at Visit 9/Month 6 or at early discontinuation) was performed for all patients. All patients who completed the assessments over the initial 6 months of the trial were eligible to continue in an additional 6-month, double-blind, placebo- controlled extension, designed to collect information on the longer-term safety and efficacy of the trial treatments.

Following completion of the 6-month Initial Treatment Period, patients that met all entry criteria were re-randomized and treated as follows:

* Patients originally randomized to one of the two dose levels of EryDex (low dose or high dose; Groups 1 or 2) continued in the same treatment arm.
* Patients originally randomized to the Placebo group (Group 3) were re-allocated as defined at the initial randomization in equal proportions (1:1) and received either the EryDex low dose or high dose as follows:

  * Following 6 months of treatment, one third of the placebo patients were switched to treatment with EryDex, as described above.
  * After 9 months of treatment, another third of the placebo patients were switched to treatment with EryDex, as described above.
  * At 12 months, all remaining placebo patients were eligible to switch to open-label treatment with EryDex, as described above.

ELIGIBILITY:
Inclusion Criteria:

1. Patient met clinical criteria for diagnosis of A-T. The neurological signs of A-T (incoordination of the head and eyes in lateral gaze deflection, gait ataxia associated with an inappropriately narrow base) must have been documented. Such signs of A-T illustrated the body systems in which changes were confirmed, but the listed changes were examples and other changes in those systems may have been observed and documented to confirm the diagnosis of A-T.
2. Patient was in autonomous gait or was helped by periodic use of a support (i.e., score for Item 1 of the full ICARS - Walking Capacities between 0 and 4, included).
3. Patient was investigated for the proven genetic diagnosis of A-T (prior documentation or by central laboratory test report).
4. Patient was at least 6 years of age.
5. Body weight was >15 kg.
6. The patient and parent/caregiver (if below the age of consent), or a legal representative, provided written informed consent to participate. If consent was provided solely by the caregiver in accordance with local regulations, the patient must have provided assent to participate in the study.

Exclusion criteria

General

1. Females that were:

   1. Pregnant or breast-feeding (for European Union [EU] countries only).
   2. Of childbearing potential, pregnant, or breast-feeding (for US and Rest of World countries) not using adequate birth control, as determined by their Healthcare Provider.
2. A disability that may have prevented the patient from completing all study requirements.
3. Current participation in another clinical study.

   Medical History and Current Status
4. Cluster differential 4 positive (CD4+) lymphocytes count <400/mm3 (for patients 6 years of age) or <150/mm3 (for patients >6 years). In presence of oral infections, like oral candidiasis, documented at the screening or recurrent as per medical history documentation, the limit increased to <200/mm3 (for patients >6 years).
5. Loss/removal of 250 mL or more of blood within the past 4 weeks prior to screening.
6. Current neoplastic disease or previous neoplastic disease not in remission for at least 2 years.
7. History of severe impairment of the immunological system.
8. Severe or unstable pulmonary disease.
9. Uncontrolled diabetes.
10. Any other severe, unstable, or serious disease or condition that in the Investigator's opinion put the patient at risk for imminent life-threatening morbidity, need for hospitalization, or mortality.
11. Any clinically significant abnormality on standard laboratory examinations (hematology, biochemistry, urinalysis) at screening that remains abnormal on repeat testing. Eligibility of patients with abnormal laboratory test values was determined by the Investigator in consultation with the Medical Monitor.
12. Confirmed hemoglobinopathies, e.g., hemoglobin C disease, sickle cell anemia, or thalassemia.
13. Moderate or severe renal and/or hepatic impairment.

    Prior/Concomitant Medication
14. Any previous oral or parenteral steroid use within 4 weeks before Baseline. Treatment with inhaled or intranasal steroids for asthma or allergies, as well as use of topical steroids will be permitted.
15. Chronic condition or prior allergic reaction representing a contraindication to the use of dexamethasone or other steroid drugs.
16. Has participated in any other trial with an investigational drug and received a dose within 30 days or 10 half-lives (whichever is greater) from the start of the 30-day Screening Period.
17. Has participated in a previous trial with EryDex.
18. Requires any concomitant medication prohibited by the protocol.
19. Has taken a drug or treatment known to cause major organ system toxicity during the past year.
20. Used of any drug that is a strong inducer/inhibitor of cytochrome P450 3A4 (CYP3A4) within 4 weeks before baseline.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guenter R. Janhofer, MD, PhD, Study Director — EryDel S.p.A
Locations (22):
- United States (4):
  - UCLA-Ataxia Center and HD Center of Exellence, Los Angeles, California
  - The Ataxia-Telangiectasia Clinical Center, The Johns Hopkins Hospital, Baltimore, Maryland
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - UT Health, Houston, Texas
- Royal Children's Hospital, Melbourne, Victoria, Australia
- Laboratoriumgeneeskunde, Leuven, Belgium
- Klinik für Kinder- und Jugendmedizin Pädiatrische Allergologie, Pneumologie und Mukoviszidose, Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse, Germany
- India (7):
  - National Institute of Mental Health and Neurosciences, Bangalore, Karnataka
  - Amrita Institute of Medical Sciences and Research Centre, Kochi, Kerala
  - Jaslok Hospital and Research Centre, Mumbai, Maharashtra
  - PD Hinduja National Hospital and Medical Research, Mahīm, Mumbai
  - Vijaya Health Centre, Department of Neurology, Chennai, Tamil Nadu
  - Nizam's Institute of Medical Sciences, Hyderabad, Telangana
  - All India Institute of Medical Sciences, New Delhi
- Sheba Medical Center, Tel Litwinsky, Israel
- Italy (2):
  - U.O. Neurologia e Psichiatria dell'Infanzia e dell' Adolescenza. ASST Spedali Civili, Piazzale Spedali Civili, 1, Brescia
  - Dipartimento di Pediatria e Neuropsichiatria Infantile, Università Sapienza di Roma, Azienda Policlinico Universitario Umberto I, Rome
- Norwegian National Unit for Newborn Screening, Division of Pediatric and Adolescent Medicine, Oslo University Hospital, Oslo, Norway
- Department of Clinical Immunology The Children's Memorial Health Institute, Warsaw, Poland
- Hospital Universitario La Paz., Madrid, Spain
- El Razi Hospital, Manouba, Tunisia
- Nottingham University Hospitals NHS Trust - Queen's Medical Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koenig MK, Leuzzi V, Gouider R, Yiu EM, Pietrucha B, Stray-Pedersen A, Perlman SL, Wu S, Burgers T, Borgohain R, Kandadai RM, Meyts I, Bucciol G, Udwadia-Hegde A, Yadav R, Roberts D, Dane A, Roden M, Thye D, Horn B, Lederman HM, Whitehouse WP. Long-term safety of dexamethasone sodium phosphate encapsulated in autologous erythrocytes in pediatric patients with ataxia telangiectasia. Front Neurol. 2025 Jan 23;15:1526914. doi: 10.3389/fneur.2024.1526914. eCollection 2024. PMID 39917433
- [Derived] Zielen S, Crawford T, Benatti L, Magnani M, Kieslich M, Ryan M, Meyts I, Gulati S, Borgohain R, Yadav R, Pal P, Hegde A, Kumar S, Venkateswar A, Udani V, Vinayan KP, Nissenkorn A, Fazzi E, Leuzzi V, Stray-Pedersen A, Pietrucha B, Pascual SI, Gouider R, Koenig MK, Wu S, Perlman S, Thye D, Janhofer G, Horn B, Whitehouse W, Lederman H. Safety and efficacy of intra-erythrocyte dexamethasone sodium phosphate in children with ataxia telangiectasia (ATTeST): a multicentre, randomised, double-blind, placebo-controlled phase 3 trial. Lancet Neurol. 2024 Sep;23(9):871-882. doi: 10.1016/S1474-4422(24)00220-5. PMID 39152028

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 176 patients were randomized, and 175 patients received study drug (Safety Population or ITT).
  There were 164 patients in the mITT and 107 patients in the PP population. Of the 164 patients in the mITT, 54 were randomized to placebo, 56 to low dose, and 54 to high dose EryDex.The PP population excluded 57 patients that were unable to comply with the study treatment interval, mainly due to the COVID-19 pandemic and issues with traveling in India, and who did not meet the definition of the PP.
Groups:
- EryDex Low Dose DSP - SAF: EDS-EP dose range of ~5-10 mg DSP/infusion: Patients were treated with EryDex prepared using 2.0 mL of the 25 mg/mL DSP solution, plus 11 mL sterile water for injection in the same syringe, for a total of 13.0 mL, corresponding to 50.0 mg of experimental drug which resulted in a mean of 8.23 mg ± 3.30 mg (mean ± standard deviation) of DSP infused to subjects. This study treatment was to be administered by IV infusion once per month for 12 consecutive months (6 months Initial Treatment Period + 6 months Extension Treatment Period). Each patient underwent a 30-day Screening Period, during which any previous treatments with other corticosteroid compounds were withdrawn (washout from previous treatment).
  Other Names:
  EryDex System end product Low dose DSP
  EryDex Low dose DSP: EDS-EP dose range of ~5-10 mg DSP/infusion
- EryDex High Dose DSP - SAF: EDS-EP dose range of ~14-22 mg DSP/infusion: Patients were treated with EryDex prepared using 5.0 mL of the 25 mg/mL DSP solution, plus 11 mL sterile water for injection in the same syringe, for a total of 16 mL, corresponding to 125 mg of experimental drug which resulted in a mean of 17.4 ± 5.38 mg (mean ± standard deviation) of DSP infused to subjects. This study treatment was to be administered by IV infusion once per month for 12 consecutive months (6 months Initial Treatment Period + 6 months Extension Treatment Period).Each patient underwent a 30-day Screening Period, during which any previous treatments with other corticosteroid compounds were withdrawn (washout from previous treatment).
  Other Names:
  EryDex System end product High dose DSP
  EryDex High dose DSP: EDS-EP dose range of ~14-22 mg DSP/infusion
- Pooled Placebo - SAF: Patients were treated with autologous erythrocytes prepared with the EDS process using a placebo solution (5 mL of 0.372% NaCl solution) instead of experimental drug (DSP). Placebo was diluted with 11 mL sterile water for injection in the same syringe, for a total of 16 mL.
  This study treatment was to be administered by IV infusion once per month for 12 consecutive months (6 months Initial Treatment Period + 6 months Extension Treatment Period).
  Each patient underwent a 30-day Screening Period, during which any previous treatments with other corticosteroid compounds were withdrawn (washout from previous treatment).
  Pooled Placebo: EDS processed autologous erythrocytes using 5 mL of 0.372% sodium chloride [NaCl] solution.
Period: Overall Study
Arm/Group | EryDex Low Dose DSP - SAF | EryDex High Dose DSP - SAF | Pooled Placebo - SAF
Started (patients randomized) | 59 | 58 | 59
Participants Who Took the Study Drug | 59 | 57 | 59
Modified Intention to Treat Population - mITT | 56 | 54 | 54
Safety Population - SAF | 59 | 57 | 59
Per Protocol Population - PP | 36 | 38 | 33
Completed Visit 9 | 43 | 46 | 43
Discontinued Prior to Visit 9 | 16 | 11 | 16
Participants From Month 6 to Month 9 | 43 | 46 | 43
Participants From Month 9 to month12 | 34 | 38 | 36
Completed | 34 | 38 | 36
Not Completed | 25 | 20 | 23
Not completed — Adverse Event | 3 | 3 | 1
Not completed — Withdrawal by Subject | 7 | 3 | 4
Not completed — Other | 0 | 1 | 0
Not completed — Covid-Related Treatment/Visit Delay | 15 | 13 | 17
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety (SAF): all patients who received any amount of randomized treatment (also referred to as the ITT ) Full Analysis Set (FAS): All randomized pts who received at least 1 dose of study medication and had at least one post-baseline efficacy assessment of the primary efficacy variable (also referred to as mITT ) Per Protocol (PP): all pts enrolled fulfilled all Inclusion/Exclusion criteria, did not have any major protocol violations, and completed the Initial Treatment Period of the study
Groups:
- Total: Total of all reporting groups
Arm/Group | EryDex Low Dose DSP - SAF | EryDex High Dose DSP - SAF | Pooled Placebo - SAF | Total
Number analyzed (Participants) | 59 | 57 | 59 | 175
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 59 | 57 | 59 | 175
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.5 (3.16) | 10.2 (4.86) | 10.3 (4.02) | 10.0 (4.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 29 | 85
  Male | 30 | 30 | 30 | 90
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 25 | 20 | 27 | 72
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3
  White | 34 | 36 | 29 | 99
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 1 | 2 | 0 | 3
  United States | 11 | 12 | 10 | 32
  Norway | 2 | 2 | 1 | 5
  Poland | 3 | 5 | 3 | 11
  United Kingdom | 2 | 3 | 6 | 11
  Italy | 1 | 2 | 1 | 4
  Israel | 1 | 0 | 0 | 1
  Australia | 1 | 3 | 1 | 5
  Tunisia | 3 | 3 | 2 | 8
  Germany | 5 | 6 | 5 | 16
  Spain | 7 | 2 | 4 | 13
  India | 22 | 18 | 26 | 66

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Modified International Cooperative Ataxia Rating Scale (mICARS)
Description: The International Cooperative Ataxia Rating Scale (ICARS) was an assessment of the degree of impairment in patients with cerebellar ataxia and was administered in its entirety; however, the primary efficacy assessment was based on the modified (m)ICARS, which excluded the Oculomotor domain (items 17 to 19) and items 8 to 12 of the Kinetic Functions domain of the ICARS.
  The mICARS was a 54 points maximum score (min 0) questionnaire divided into 3 sections:
  * Posture and Gait Disturbance section-7 items (min score 0, max score 34)
  * Kinetic Function-2 items (min score 0, max score 12)
  * Speech Disorder- 2 items (min score 0, max score 8). The assessment was designed to be completed within 30 minutes, and higher scores - both for total and subscores - indicate a higher level of disease impairment. The subscores are added to give the total score.
Time Frame: to Month 6 (Visit 9)
Population: Modified Intention to Treat population - mITT: ll randomized patients who received at least one dose of study medication and had at least one post-baseline efficacy assessment of the primary efficacy variable
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- EryDex Low Dose DSP - mITT: EDS-EP dose range of ~5-10 mg DSP/infusion. This study treatment was to be administered by IV infusion once per month for 12 consecutive months (6 months Initial Treatment Period + 6 months Extension Treatment Period). Each patient underwent a 30-day Screening Period, during which any previous treatments with other corticosteroid compounds were withdrawn (washout from previous treatment).
  Other Names:
  EryDex System end product Low dose DSP
  EryDex Low dose DSP: EDS-EP dose range of ~5-10 mg DSP/infusion
- EryDex High Dose DSP - mITT: EDS-EP dose range of ~14-22 mg DSP/infusion. This study treatment was to be administered by IV infusion once per month for 12 consecutive months (6 months Initial Treatment Period + 6 months Extension Treatment Period).Each patient underwent a 30-day Screening Period, during which any previous treatments with other corticosteroid compounds were withdrawn (washout from previous treatment).
  Other Names:
  EryDex System end product High dose DSP
  EryDex High dose DSP: EDS-EP dose range of ~14-22 mg DSP/infusion
- Placebo - mITT: Patients were treated with autologous erythrocytes prepared with the EDS process using a placebo solution (NaCl solution) instead of experimental drug (DSP).
  This study treatment was to be administered by IV infusion once per month for 12 consecutive months (6 months Initial Treatment Period + 6 months Extension Treatment Period).
  Each patient underwent a 30-day Screening Period, during which any previous treatments with other corticosteroid compounds were withdrawn (washout from previous treatment).
  Pooled Placebo: EDS processed autologous erythrocytes using 5 mL of 0.372% sodium chloride [NaCl] solution.
Arm/Group | EryDex Low Dose DSP - mITT | EryDex High Dose DSP - mITT | Placebo - mITT
Number analyzed (Participants) | 56 | 54 | 54
score on a scale | 0.8 (3.56) | 1.0 (3.32) | 2.3 (5.03)
Statistical Analysis 1: Comparison: EryDex Low Dose DSP - mITT vs Placebo - mITT; Least squares means, and p-values are derived from a mixed model repeated measures analysis with baseline modified ICARS value as covariate and the fixed effects of treatment, age, sex, region and visit and the interaction term treatment-by-visit; Test type: Superiority; p = 0.0847, Mixed model for repeated measures; Least squares mean difference = -1.37, 95% CI 2-sided [-2.932 to 0.190]
Statistical Analysis 2: Comparison: EryDex High Dose DSP - mITT vs Placebo - mITT; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0765, Mixed model for repeated measures; Least squares mean difference = -1.40, 95% CI 2-sided [-2.957 to 0.152]

2. Secondary Outcome: Number of Patients With Improving, Stable or Worsening Score Using a Clinical Global Impression of Change (CGI-C)
Description: The CGI-C scale assesses the change in the patient's clinical status from baseline using a 7-point scale, ranging from 1 (very much improved) to 7 (very much worse), with a score of 4 indicating no change. Clinicians were required to conduct a full clinical interview and examination of the patient.
  The interview and examination assessed various aspects of the patient's appearance (grooming, evidence of falls, etc.), ataxia, cognition (orientation, calculation ability, language, ability to follow commands, memory, etc.), apraxia, dysarthria, extrapyramidal motor symptoms, activities of daily living, and mood. The higher the score the worse the outcome.
Time Frame: to Month 6 (Visit 9)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- EryDex High Dose DSP - mITT: EDS-EP dose range of ~14-22 mg DSP/infusion. This study treatment was to be administered by IV infusion once per month for 12 consecutive months (6 months Initial Treatment Period + 6 months Extension Treatment Period). Each patient underwent a 30-day Screening Period, during which any previous treatments with other corticosteroid compounds were withdrawn (washout from previous treatment).
  Other Names:
  EryDex System end product High dose DSP
  EryDex High dose DSP: EDS-EP dose range of ~14-22 mg DSP/infusion
Arm/Group | EryDex Low Dose DSP - mITT | EryDex High Dose DSP - mITT | Placebo - mITT
Number analyzed (Participants) | 56 | 54 | 54
Participants
  Improvement (Scores 1-3) | 19 | 27 | 19
  Stable or Worsening (Scores 4-7) | 37 | 27 | 35
Statistical Analysis 1: Comparison: EryDex Low Dose DSP - mITT vs Placebo - mITT; Logistic regression modeling (0/1), where 0 = No change or worsening and 1= improvement, with age (at 2 levels: <10 years, ≥10 years), sex, treatment, region as fixed effects; Test type: Superiority; p = 0.8919, Regression, Logistic; Odds Ratio (OR) = 0.946, 95% CI 2-sided [0.426 to 2.099]
Statistical Analysis 2: Comparison: EryDex High Dose DSP - mITT vs Placebo - mITT; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1255, Regression, Logistic; Odds Ratio (OR) = 1.848, 95% CI 2-sided [0.842 to 4.053]

3. Secondary Outcome: Number of Patients With None to Severe (0 to 4) Scores in Clinical Global Impression of Severity (CGI-S)-Structured of Neurological Symptoms of AT
Description: The CGI-S scale measures global severity of illness at a given point in time, and is usually rated on a 7-point, Likert-type scale ranging from 1 (normal, not ill at all) to 7 (among the most extremely ill patients). No version of the CGI-S exists which has been specifically adapted for use in patients with A-T; therefore, a 5-point version was developed that considered the severity of the following symptoms of A-T: ataxia (walking), dysarthria, dysmetria, extrapyramidal symptoms (chorea, myoclonus, dystonia, and tremor), and eye movements. Ratings of none (0), mild (1), moderate (2), severe (3), and very severe (4) were selected based on the level of symptomatology. The higher the score the worse the outcome.
Time Frame: to Visit 9 (Month 6)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | EryDex Low Dose DSP - mITT | EryDex High Dose DSP - mITT | Placebo - mITT
Number analyzed (Participants) | 56 | 54 | 54
Participants
  CGI-S Score - 0 | 0 | 0 | 0
  CGI-S Score - 1 | 15 | 16 | 17
  CGI-S Score - 2 | 29 | 26 | 24
  CGI-S Score - 3 | 12 | 12 | 13
  CGI-S Score - 4 | 0 | 0 | 0
Statistical Analysis 1: Comparison: EryDex Low Dose DSP - mITT vs Placebo - mITT; Odds ratio, confidence limits, and p-value derived using a proportional odds ordinal logistic regression analysis, with age (at 2 levels: <10 years, ≥10 years), sex, treatment, region, visit, baseline CGI-S score, and treatment-by- visit interaction as fixed effects; Test type: Superiority; p = 0.4583, Ordinal Logistic Regression Analysis; Odds Ratio (OR) = 1.369, 95% CI 2-sided [0.597 to 3.144]
Statistical Analysis 2: Comparison: EryDex High Dose DSP - mITT vs Placebo - mITT; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.4585, Ordinal Logistic Regression Analysis; Odds Ratio (OR) = 1.371, 95% CI 2-sided [0.595 to 3.160]

4. Secondary Outcome: Change From Baseline of Vineland Adaptive Behavior Scale (VABS-II) Scores - Last Observation Carried Forward (LOCF)
Description: VABS-II was a questionnaire to assess adaptive behavior. It contained 4 domains each with 2-3 subdomains, every subdomain contained various items (questions):
  A) communication (receptive, expressive, written) B) daily living skills (personal, domestic, community) C) socialization (interpersonal relationships, play and leisure time, coping skills) D) motor skills (gross motor, fine motor). The expanded version of the VABS consisted of 540 items, 261 of which used in this trial.
  The possible score for each item was from 0 to 4 based on whether the patient performed the activity "never", "rarely", "sometimes", "often" or "almost always".
  At the end of each domain section, a total score (the sum of the score for each item) was calculated. Domain A: min score 0, max score 572. Domain B: 0 - 800. Domain C: 0 - 580. Domain D: 0 - 424. A grand total score (A+B+C+D scores) was provided (range:0-2376) The lower the score the higher the disability at each level (domains and subdomains).
Time Frame: to Visit 9 (Month 6)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EryDex Low Dose DSP - mITT | EryDex High Dose DSP - mITT | Placebo - mITT
Number analyzed (Participants) | 56 | 52 | 52
score on a scale | 42.6 (125.95) | -26.5 (214.52) | 57.5 (200.37)
Statistical Analysis 1: Comparison: EryDex Low Dose DSP - mITT vs Placebo - mITT; Least squares means difference, associated statistics, and p-values derived using ANCOVA, with age (at 2 levels: <10 years, >=10 years), sex, treatment, region, and baseline VABS score as fixed effects; Test type: Superiority; p = 0.7029, ANCOVA; Least squares means difference = -13.33, 95% CI 2-sided [-82.261 to 55.601]
Statistical Analysis 2: Comparison: EryDex High Dose DSP - mITT vs Placebo - mITT; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0328, ANCOVA; Least squares means difference = -77.31, 95% CI 2-sided [-148.201 to -6.421]

5. Secondary Outcome: Number of Patients With at Least One Treatment-Emergent Adverse Event (TEAE) at Month 6
Description: TEAE = Treatment Emergent Adverse Events were any AEs started on or after the day of the first infusion through the day just prior to the day of the Visit 9 ("Month 6") infusion, or <=60 days after last dose if the subject never continued past this period.
Time Frame: to Visit 9 (Month 6)
Population: Safety Population (SAF): all patients who received any amount of randomized treatment (also referred to as the ITT population).
Measure: Count of Participants; unit: Participants
Groups:
- EryDex Low Dose DSP - SAF: EDS-EP dose range of ~5-10 mg DSP/infusion. This study treatment was to be administered by IV infusion once per month for 12 consecutive months (6 months Initial Treatment Period + 6 months Extension Treatment Period). Each patient underwent a 30-day Screening Period, during which any previous treatments with other corticosteroid compounds were withdrawn (washout from previous treatment).
  Other Names:
  EryDex System end product Low dose DSP
  EryDex Low dose DSP: EDS-EP dose range of ~5-10 mg DSP/infusion
- EryDex High Dose DSP - SAF: EDS-EP dose range of ~14-22 mg DSP/infusion. This study treatment was to be administered by IV infusion once per month for 12 consecutive months (6 months Initial Treatment Period + 6 months Extension Treatment Period).Each patient underwent a 30-day Screening Period, during which any previous treatments with other corticosteroid compounds were withdrawn (washout from previous treatment).
  Other Names:
  EryDex System end product High dose DSP
  EryDex High dose DSP: EDS-EP dose range of ~14-22 mg DSP/infusion
- Pooled Placebo - SAF: Patients were treated with autologous erythrocytes prepared with the EDS process using a placebo solution (NaCl solution) instead of experimental drug (DSP).
  This study treatment was to be administered by IV infusion once per month for 12 consecutive months (6 months Initial Treatment Period + 6 months Extension Treatment Period).
  Each patient underwent a 30-day Screening Period, during which any previous treatments with other corticosteroid compounds were withdrawn (washout from previous treatment).
  Pooled Placebo: EDS processed autologous erythrocytes using 5 mL of 0.372% sodium chloride [NaCl] solution.
Arm/Group | EryDex Low Dose DSP - SAF | EryDex High Dose DSP - SAF | Pooled Placebo - SAF
Number analyzed (Participants) | 59 | 57 | 59
Participants
  Patients With Pre- treatment AE | 14 | 16 | 14
  Patients With Any TEAE | 43 | 47 | 43
  Patients With Any Treatment-related TEAE | 15 | 21 | 15
  Patients With Any Serious TEAE | 6 | 7 | 7
  Patients With Any Serious Treatment-related TEAE | 0 | 1 | 0
  Patients With Any TEAE Leading to Discontinuation | 0 | 2 | 0
  Patients With Any TEAE Leading to Death | 0 | 0 | 0

6. Secondary Outcome: Number of Patients With at Least One Treatment-Emergent Adverse Event (TEAE) at Month 12
Description: TEAE = Treatment Emergent Adverse Events were any AEs started on or after the day of the first infusion through the day just prior to the day of the Visit 15 ("Month 12") infusion.
  Placebo patients who switched to EryDex treatment at 6 and 9 months were not added to the Extension Treatment Period safety data so that the results reported here under are for those patients who remained on placebo from the start of the study till the end of it.
Time Frame: to Visit 15 (Month 12)
Population: Safety Population: all patients who received any amount of randomized treatment (also referred to as the ITT population). Placebo patients who switched to EryDex treatment at 6 and 9 months were not added to the Extension Treatment Period safety data so that the results reported are for those patients who remained on placebo from the start of the study (N=19)
Measure: Count of Participants; unit: Participants
Groups:
- EryDex High Dose DSP - SAF: EDS-EP dose range of ~14-22 mg DSP/infusion. This study treatment was to be administered by IV infusion once per month for 12 consecutive months (6 months Initial Treatment Period + 6 months Extension Treatment Period). Each patient underwent a 30-day Screening Period, during which any previous treatments with other corticosteroid compounds were withdrawn (washout from previous treatment).
  Other Names:
  EryDex System end product High dose DSP
  EryDex High dose DSP: EDS-EP dose range of ~14-22 mg DSP/infusion
- Non-switch Placebo - SAF: Patients were treated with autologous erythrocytes prepared with the EDS process using a placebo solution (NaCl solution) instead of experimental drug (DSP).
  This study treatment was to be administered by IV infusion once per month for 12 consecutive months (6 months Initial Treatment Period + 6 months Extension Treatment Period).
  Each patient underwent a 30-day Screening Period, during which any previous treatments with other corticosteroid compounds were withdrawn (washout from previous treatment).
  Pooled Placebo: EDS processed autologous erythrocytes using 5 mL of 0.372% sodium chloride [NaCl] solution.
Arm/Group | EryDex Low Dose DSP - SAF | EryDex High Dose DSP - SAF | Non-switch Placebo - SAF
Number analyzed (Participants) | 59 | 57 | 19
Participants
  Patients With Any TEAE | 45 | 50 | 15
  Patients With Any Treatment-related TEAE | 19 | 25 | 5
  Patients With Any Serious TEAE | 8 | 9 | 4
  Patients With Any Serious Treatment-related TEAE | 1 | 1 | 1
  Patients With Any TEAE Leading to Discontinuation | 1 | 2 | 0
  Patients With Any TEAE Leading to Death | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: TEAEs were all the AEs reported up to the end of the Extension Treatment Period (Month 12). All AEs with an onset date on/after the start of the first infusion through 60 days after the last dose are included. A patient with more than one event with the same SOC is counted once
Description: Only AEs in the these arms/groups of interest were calculated: EryDex low dose and high dose, non-switch placebo, placebo patients who switched to EryDex (low dose or high dose) at 6 and 9 months, and patients remained on placebo till the end of the study. Please note that data collected on "placebo pre switch" group corresponds to data reported for placebo patients in the 6-Month Initial Treatment Period.
Groups:
- Non-switch Placebo - SAF: Patients were treated with autologous erythrocytes prepared with the EDS process using a placebo solution (5 mL of 0.372% NaCl solution) instead of experimental drug (DSP). Placebo was diluted with 11 mL sterile water for injection in the same syringe, for a total of 16 mL.
  This study treatment was to be administered by IV infusion once per month for 12 consecutive months (6 months Initial Treatment Period + 6 months Extension Treatment Period).
  Each patient underwent a 30-day Screening Period, during which any previous treatments with other corticosteroid compounds were withdrawn (washout from previous treatment).
  Pooled Placebo: EDS processed autologous erythrocytes using 5 mL of 0.372% sodium chloride [NaCl] solution.
- Placebo Patients Switch to Low Dose - Month 6: Patients originally randomized to the Placebo group (Pooled Placebo) re-allocated in EryDex low dose at Month 6 - Visit 9. (N=9)
- Placebo Patients Switch to High Dose - Month 6: Patients originally randomized to the Placebo group (Pooled Placebo) re-allocated in EryDex High dose at Month 6 - Visit 9. (N=9)
- Placebo Patients Switch to Low Dose - Month 9: Patients originally randomized to the Placebo group (Pooled Placebo) re-allocated in EryDex low dose at Month 9 - Visit 12 . (N=11)
- Placebo Patients Switch to High Dose - Month 9: Patients originally randomized to the Placebo group (Pooled Placebo) re-allocated in EryDex low dose at Month 9 - Visit 12. (N=11)
Arm/Group | EryDex Low Dose DSP - SAF | EryDex High Dose DSP - SAF | Non-switch Placebo - SAF | Placebo Patients Switch to Low Dose - Month 6 | Placebo Patients Switch to High Dose - Month 6 | Placebo Patients Switch to Low Dose - Month 9 | Placebo Patients Switch to High Dose - Month 9
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/57 | 1/19 | 0/9 | 0/9 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 8/59 | 9/57 | 4/19 | 1/9 | 1/9 | 1/11 | 4/11
Other Adverse Events (participants affected / at risk) | 45/59 | 50/57 | 15/19 | 7/9 | 8/9 | 7/11 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EryDex Low Dose DSP - SAF (N=59) | EryDex High Dose DSP - SAF (N=57) | Non-switch Placebo - SAF (N=19) | Placebo Patients Switch to Low Dose - Month 6 (N=9) | Placebo Patients Switch to High Dose - Month 6 (N=9) | Placebo Patients Switch to Low Dose - Month 9 (N=11) | Placebo Patients Switch to High Dose - Month 9 (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepato-Lenticular Degeneration (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Herpes Zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacterial test positive (Investigations) | 4 | 6 | 3 | 1 | 0 | 1 | 2
Juvenile idiophatic arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
B-cell limphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dystonia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EryDex Low Dose DSP - SAF (N=59) | EryDex High Dose DSP - SAF (N=57) | Non-switch Placebo - SAF (N=19) | Placebo Patients Switch to Low Dose - Month 6 (N=9) | Placebo Patients Switch to High Dose - Month 6 (N=9) | Placebo Patients Switch to Low Dose - Month 9 (N=11) | Placebo Patients Switch to High Dose - Month 9 (N=11)
Anemia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hepato-lenticular degeneration (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Talipes (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tympanic membrane scarring (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Astigmatism (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye movement disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Papilloedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 4 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal prurirus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 6 | 5 | 0 | 0 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 4 | 0 | 1 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Teething (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 13 | 11 | 3 | 0 | 1 | 1 | 2
Catheter site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Extravasation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 3 | 0 | 0 | 0 | 1 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 15 | 19 | 3 | 3 | 2 | 4 | 2
Swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 4 | 2 | 1 | 1 | 1 | 0 | 0
Conjuntivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 5 | 2 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 4 | 1 | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Molluscum contagiosum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 10 | 11 | 5 | 1 | 1 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 3 | 0 | 1 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 9 | 1 | 1 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 1 | 0 | 1 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacterial test positive (Investigations) | 10 | 10 | 4 | 1 | 2 | 1 | 3
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood iron decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Blood lactate dehidrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bone density decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest expansion decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Low density lipoprotein increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Platelet count increased (Investigations) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Respiratory rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 2 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertrygliceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Insulin resistance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 6 | 5 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal stifness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 2
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Decreased vibratory sense (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Dystonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 8 | 5 | 2 | 2 | 0 | 1 | 2
Lethargy (Nervous system disorders) | 1 | 3 | 0 | 1 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Parkinsonism (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pineal gland cyst (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Affect lability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Emotional poverty (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enuresis (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 3 | 0 | 1 | 1 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysmenerrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 13 | 6 | 1 | 4 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 3 | 0 | 1 | 2 | 1
Acanthosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 0
Granuloma skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 10 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT02770807/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT02770807/SAP_001.pdf